CLINICAL TRIAL: NCT06307223
Title: Efficacy and Safety of 30% Supramolecular Salicylic Acid Combined With Supramolecular Active Zinc in the Treatment of Malassezia Folliculitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240301
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Malassezia Folliculitis
Keywords: malassezia folliculitis; supramolecular salicylic acid; zinc pyrithione; clinical research; treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30% supramolecular salicylic acid combined with supramolecular active zinc treatment group (Experimental): The patients received weekly application of 30% supramolecular salicylic acid in conjunction with daily application of topical supramolecular active zinc anti-dandruff lotion, for a duration of 8 weeks.
  Interventions: Drug: 30% supramolecular salicylic acid; Drug: supramolecular active zinc

INTERVENTIONS:
Drug: 30% supramolecular salicylic acid — The patients received weekly application of 30% supramolecular salicylic acid for a duration of 8 weeks.
Drug: supramolecular active zinc — The patients received daily application of topical supramolecular active zinc anti-dandruff lotion for a duration of 8 weeks.

SUMMARY:
Malassezia folliculitis is a common dermatological disorder. While antifungal agents generally demonstrate efficacy in application, the prevalence of recurrence and drug resistance remains a common occurrence. Supramolecular salicylic acid represents a novel class of superficial chemical peel agents, exhibiting keratolytic, anti-inflammatory, and bacteriostatic properties. Zinc pyrithione has broad spectrum antibacterial, antifungal, and anti-inflammatory effects. In the present study, investigators evaluated the clinical efficacy of topical application of supramolecular salicylic acid in combination with zinc pyrithione for the treatment and prevention of Malassezia folliculitis recurrence. All data are recorded and compared after the end of the experiment. The enrolled patients received daily application of topical supramolecular active zinc anti-dandruff lotion, in conjunction with weekly application of 30% supramolecular salicylic acid, for a duration of 8 weeks. Lesion counts, Malassezia detection, clinical symptom scores, patient satisfaction, and side effects were recorded at each visit till the week 12.

DETAILED DESCRIPTION:
Malassezia folliculitis is a common dermatological disorder. While antifungal agents generally demonstrate efficacy in application, the prevalence of recurrence and drug resistance remains a common occurrence. Supramolecular salicylic acid represents a novel class of superficial chemical peel agents, exhibiting keratolytic, anti-inflammatory, and bacteriostatic properties. Zinc pyrithione has broad spectrum antibacterial, antifungal, and anti-inflammatory effects. In the present study, investigators evaluated the clinical efficacy of topical application of supramolecular salicylic acid in combination with zinc pyrithione for the treatment and prevention of Malassezia folliculitis recurrence. The enrolled patients received daily application of topical supramolecular active zinc anti-dandruff lotion, in conjunction with weekly application of 30% supramolecular salicylic acid, for a duration of 8 weeks. Lesion counts, Malassezia detection, clinical symptom scores, patient satisfaction, and side effects were recorded at each visit till the week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females, aged 18-65 years old;
2. Diagnosed as Malassezia folliculitis;
3. The total lesion counts of the anterior chest or posterior dorsal skin ranged from 30 to 100 (included papules, pustules, and papulopustules).

Exclusion Criteria:

1. Suffering other skin diseases that may influence the result;
2. Established allergy to supramolecular salicylic acid or supramolecular active zinc;
3. Pregnant and lactating patients;
4. Patients who had received oral antifungal treatment within 4 months before the trial (or topical antifungal treatment within 2 months); had received oral antibiotics, glucocorticoids, and other folliculitis drugs within 4 weeks; or used physiotherapy for folliculitis; or treated with salicylic acid and alpha hydroxy acid; or used other topical medications for folliculitis within 2 weeks;
5. History of injection or surgery at the affected site within 2 months before the trial;
6. Immunodeficiency diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
lesion counts | From enrollment to week 12
  The counts of skin lesions, including papules, pustules, and papulopustules.
The reduction rate of lesion counts | From week 1 to week 12
  The reduction rate expressed as (lesion counts at baseline - lesion counts at 8 weeks)/lesion counts at baseline×100%.
Clinical efficacy | week 8 and week 12
  The clinical efficacy after the treatment was classified as follows: clinical cure (refers to lesion reduction rate of 100%, negative Malassezia detection), obvious improvement (refers to lesion reduction rate of 70-99%, positive or negative Malassezia detection), moderate improvement (refers to lesion reduction rate of 30-69%, positive or negative Malassezia detection), and no improvement (refers to lesion reduction rate <30%, positive Malassezia detection).

SECONDARY OUTCOMES:
Clinical symptoms scores | From enrollment to week 12
  The degree of clinical symptoms, including pruritus, scale, greasiness, and erythema, was classified as 0 (none), 2 (mild), 4 (moderate), 6 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vlachos C, Henning MAS, Gaitanis G, Faergemann J, Saunte DM. Critical synthesis of available data in Malassezia folliculitis and a systematic review of treatments. J Eur Acad Dermatol Venereol. 2020 Aug;34(8):1672-1683. doi: 10.1111/jdv.16253. Epub 2020 Apr 30. PMID 32012377
- [Result] Roques C, Brousse S, Panizzutti C. In vitro antifungal efficacy of ciclopirox olamine alone and associated with zinc pyrithione compared to ketoconazole against Malassezia globosa and Malassezia restricta reference strains. Mycopathologia. 2006 Dec;162(6):395-400. doi: 10.1007/s11046-006-0075-0. PMID 17146583
- [Result] Berger RS, Fu JL, Smiles KA, Turner CB, Schnell BM, Werchowski KM, Lammers KM. The effects of minoxidil, 1% pyrithione zinc and a combination of both on hair density: a randomized controlled trial. Br J Dermatol. 2003 Aug;149(2):354-62. doi: 10.1046/j.1365-2133.2003.05435.x. PMID 12932243
- [Result] Park M, Cho YJ, Lee YW, Jung WH. Understanding the Mechanism of Action of the Anti-Dandruff Agent Zinc Pyrithione against Malassezia restricta. Sci Rep. 2018 Aug 14;8(1):12086. doi: 10.1038/s41598-018-30588-2. PMID 30108245
- [Result] Magerusan SE, Hancu G, Rusu A. A Comprehensive Bibliographic Review Concerning the Efficacy of Organic Acids for Chemical Peels Treating Acne Vulgaris. Molecules. 2023 Oct 22;28(20):7219. doi: 10.3390/molecules28207219. PMID 37894698
- [Result] Henning MAS, Hay R, Rodriguez-Cerdeira C, Szepietowski JC, Piraccini BM, Ferreiros MP, Arabatzis M, Sergeev A, Nenoff P, Kotrekhova L, Nowicki RJ, Faergemann J, Padovese V, Prohic A, Skerlev M, Schmid-Grendelmeier P, Sigurgeirsson B, Gaitanis G, Lecerf P, Saunte DML. Position statement: Recommendations on the diagnosis and treatment of Malassezia folliculitis. J Eur Acad Dermatol Venereol. 2023 Jul;37(7):1268-1275. doi: 10.1111/jdv.18982. Epub 2023 Mar 13. PMID 36912427
- [Result] Theelen B, Cafarchia C, Gaitanis G, Bassukas ID, Boekhout T, Dawson TL Jr. Malassezia ecology, pathophysiology, and treatment. Med Mycol. 2018 Apr 1;56(suppl_1):S10-S25. doi: 10.1093/mmy/myx134. PMID 29538738
- [Derived] Liang J, Chen Y, Yang M, Liu H, Liu Y, He S, Wang Z, Zeng W. Efficacy and safety of tranilast combined with minocycline in the treatment of moderate-to-severe rosacea: a prospective, randomized controlled study. J Dermatolog Treat. 2026 Dec;37(1):2597711. doi: 10.1080/09546634.2025.2597711. Epub 2025 Dec 22. PMID 41424372